CLINICAL TRIAL: NCT02678338
Title: A Phase I Dose Escalation Trial of the Humanized Anti-CD47 Monoclonal Antibody Hu5F9-G4 in Haematological Malignancies (CAMELLIA)
Brief Title: CAMELLIA: Anti-CD47 Antibody Therapy in Haematological Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCI-CD47-002; 2015-000720-29 (EudraCT Number)
Record Dates: First submitted 2016-01-27; First posted 2016-02-09 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — magrolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hu5F9-G4 (Experimental): Dose Escalation: CD47 blocking antibody Hu5F9-G4
  Interventions: Drug: Hu5F9-G4

INTERVENTIONS:
Drug: Hu5F9-G4

SUMMARY:
This phase I trial studies the side effects and best dose of anti-cluster of differentiation (CD)47 monoclonal antibody Hu5F9-G4 in treating patients with haematological malignancies including acute myeloid leukemia that has returned after a period of improvement (relapsed) or has not responded to previous treatment (refractory), or high risk myelodysplastic syndrome. Monoclonal antibodies, such as anti-CD47 monoclonal antibody Hu5F9-G4, block cancer growth in different ways by targeting certain cells.

ELIGIBILITY:
Key Inclusion Criteria:

* Pathologically confirmed relapsed or refractory (primary refractory and relapsed refractory) Acute Myeloid Leukemia (AML) (defined by World Health Organization (WHO) criteria) for which no further conventional therapy is suitable for the patient, or confirmed myelodysplastic syndrome defined according to WHO classification, with an International Prognostic Scoring System (IPSS) risk category of intermediate-2 or high risk, that is relapsed, refractory or intolerant to conventional therapy within 3 weeks of registration.
* Male or female, Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance score of 0-1
* Willing to undergo blood transfusions as deemed clinically necessary.
* Adequate hematological, liver, and kidney function

Key Exclusion Criteria:

* Females: Pregnant or breast-feeding women, or women of childbearing potential unless effective method of contraception is used during and for 3 months after the trial. Males: unless an effective method of contraception is used during and for 3 months after the trial.
* Any prior exposure to Hu5F9-G4 or other CD47 targeting agents.
* Treatment with any other investigational agent within 28 days prior to enrolment.
* Previous allogeneic stem cell transplant within 6 months prior to enrolment, active graft vs host disease (GVHD), or requiring transplant-related immunosuppression
* Evidence for active CNS involvement by leukaemia
* Clinical evidence or known history of cardiopulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of Hu5F9-G4, graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 (Part A) | Up to 28 days
  MTD is defined as the highest dosing schedule cohort level at which no more than 1 of 6 patients experience a Dose Limiting Toxicity (DLT).

CONTACTS AND LOCATIONS:
Overall Officials: Paresh Vyas, FRCP FRCPath, Principal Investigator — University of Oxford; Mark Chao, MD PhD, Study Director — Gilead Sciences
Locations (5):
- United Kingdom (5):
  - University Hospital of Wales, Cardiff
  - St. James University Hospital, Leeds
  - The Royal Liverpool University Hospital, Liverpool
  - The Christie NHS Foundation Trust, Manchester
  - Churchill Hospital, Oxford

REFERENCES:
- [Derived] Brierley CK, Staves J, Roberts C, Johnson H, Vyas P, Goodnough LT, Murphy MF. The effects of monoclonal anti-CD47 on RBCs, compatibility testing, and transfusion requirements in refractory acute myeloid leukemia. Transfusion. 2019 Jul;59(7):2248-2254. doi: 10.1111/trf.15397. Epub 2019 Jun 10. PMID 31183877